CLINICAL TRIAL: NCT03141255
Title: Cardiogenic Shock Intravascular Cooling Trial (CHILL-SHOCK)
Brief Title: Cardiogenic Shock Intravascular Cooling Trial
Acronym: CHILL-SHOCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: ZOLL Circulation, Inc., USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-1728
Record Dates: First submitted 2017-05-01; First posted 2017-05-05 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Cardiogenic Shock
Keywords: Therapeutic Hypothermia (TH)
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Group (No Intervention): Patients will receive only standard of care treatment for cardiogenic shock.
- Therapeutic Hypothermia (Experimental): Patients will be cooled to between 32°C and 34°C using the IVTM™ System and the Quattro® Catheter in addition to receiving standard of care treatment for cardiogenic shock.
  Interventions: Device: IVTM™ System; Device: Quattro® Catheter

INTERVENTIONS:
Device: IVTM™ System — TH will be initiated and maintained for 24 hours using the IVTM™ System and the Quattro® Catheter. After 24 hours of maintained TH, patients will be rewarmed to normal body temperature using the same Quattro® Catheter.
  Arms: Therapeutic Hypothermia
Device: Quattro® Catheter — TH will be initiated and maintained for 24 hours using the IVTM™ System and the Quattro® Catheter. After 24 hours of maintained TH, patients will be rewarmed to normal body temperature using the same Quattro® Catheter.
  Arms: Therapeutic Hypothermia

SUMMARY:
The purpose of the study is to compare patients with cardiogenic shock who receive standard therapy plus therapeutic hypothermia (TH) to patients with cardiogenic shock who receive standard medical therapy alone in order to assess the safety of TH in patients with cardiogenic shock. This study will also help understand the physiologic effects of TH in patients with cardiogenic shock. This will be a pilot study to establish the initial safety of TH and to assess tolerability of TH in this patient population.

DETAILED DESCRIPTION:
This is an unblinded pilot study of 20 patients randomized to either TH plus standard medical care or to standard medical care alone. All patients will undergo pulmonary artery (PA) catheter placement as part of the standard of care for management of cardiogenic shock. Data from the PA catheter is vital in monitoring real-time hemodynamics, initiating vasopressors/inotropes, assessing the response to the therapies, and possible need for escalation of therapy.

For patients randomized to TH, cooling to 32-34°C will then be initiated and maintained for 24 hours using the FDA-approved Intravascular Temperature Management (IVTM™) System with the 9.3 French Quattro® Catheter. The IVTM™ System along with the Quattro® Catheter are currently FDA-approved for use in cardiac surgery patients to achieve and maintain normothermia during surgery and in recovery and to induce, maintain, and reverse mild hypothermia in neurosurgery patients during surgery and in recovery. The IVTM™ System and Quattro® Catheter are not, however, currently FDA-approved to achieve therapeutic hypothermia in cardiogenic shock patients. TH is achieved by circulating normal saline in a closed system through the catheter. The temperature is measured and adjustments are made by the thermal regulation system to automatically maintain target temperature. The target temperature is achieved within 2-3 hours of initiation of TH. Rewarming is accomplished using the same balloon catheter system and heat exchange occurs without infusion of any saline or fluids.

Standard medical therapy for all patients will be based on the current recommendations for management of cardiogenic shock. This includes inotropic therapy for cardiac support, vasopressor therapy to achieve target blood pressure, diuretics for volume removal, and mechanical circulatory support as clinically indicated. Laboratory, echocardiographic, and hemodynamic parameters will be obtained for patients prior to randomization, after 18-24 hours post-randomization, and after 48-96 hours post-randomization. Core temperature will be measured via either thermal tip at the end of a transurethral urinary catheter or endotracheal temperature probe in intubated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Cardiogenic shock

   1. Systolic blood pressure <90mmHg for at least 30 minutes
   2. Cardiac Index < 2.2 L/min/m2
   3. Pulmonary capillary wedge pressure (PCWP) ≥ 15mmHg
   4. Need for central venous access, vasopressors, inotropes and/or mechanical circulatory support (i.e. intra-aortic balloon pump, Impella®, ECMO) to maintain systolic blood pressure ≥ 90mmHg
2. Etiology of shock

   1. Acute coronary syndromes (STEMI, NSTEMI, or UA)
   2. Ischemic or non-ischemic cardiomyopathy
   3. Myocarditis
   4. Hypertrophic cardiomyopathy
   5. Stress-induced cardiomyopathy
   6. Peripartum cardiomyopathy
   7. Cardiogenic shock in a patient with heart failure with preserved ejection fraction
3. Age ≥ 18 years AND ≤ 89 years
4. Admission to the University of Chicago Coronary Care Unit

Exclusion Criteria:

1. Baseline heart rate < 60 beats per minute
2. Baseline temperatures < 35°C
3. Recent cardiotomy
4. History of cardiac transplantation
5. Current pregnancy
6. Contraindication to 9.3 French femoral venous access for placement of intravascular cooling catheter
7. Hospice designation (either currently in hospice or previously enrolled within the past 30 days)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D. Paul, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Therapeutic Hypothermia
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Therapeutic Hypothermia | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 63.6 (10.3) | 62.2 (10.8) | 62.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 2.1 [1.7 to 2.4] | 2.7 [1.6 to 4.1] | 2.2 [1.7 to 3.3]
BMI (kg/mg) [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (6.8) | 30.1 (5.4) | 30.7 (6.0)
Ejection Fraction on initial "TTE" [Mean (Standard Deviation); unit: percentage of ejection fraction] — Population: Deviation from the protocol, 2/10 control patients have TTE performed at the base line.
  percentage of ejection fraction | 30.3 (14.4) | 34 (20) | 32.3 (17.4)
Admission NT-proBNP [Mean (Standard Deviation); unit: pg/mL] — Population: Deviation from the protocol, 4/10 control patients and 6/10 Therapeutic Hypothermia patients have TTE performed at the base line.
  pg/mL
    number analyzed (Participants) | 6 | 4 | 10
    (all) | 15056 (11751.4) | 29561.3 (26575.1) | 20858.1 (19189.6)
CAD [Count of Participants; unit: Participants] | 5 | 6 | 11
DM [Count of Participants; unit: Participants] | 7 | 6 | 13
HTN [Count of Participants; unit: Participants] | 10 | 10 | 20
CVA [Count of Participants; unit: Participants] | 2 | 3 | 5
Atrial fibrillation [Count of Participants; unit: Participants] | 3 | 2 | 5
Beta-blockers [Count of Participants; unit: Participants] | 9 | 7 | 16
ACEi [Count of Participants; unit: Participants] | 5 | 2 | 7
ARB [Count of Participants; unit: Participants] | 1 | 3 | 4
Neprilysin Inhibitor [Count of Participants; unit: Participants] | 1 | 2 | 3
ASA [Count of Participants; unit: Participants] | 7 | 9 | 16
Anti-platelet agent [Count of Participants; unit: Participants] | 3 | 3 | 6
Statin [Count of Participants; unit: Participants] | 8 | 7 | 15
Diuretic [Count of Participants; unit: Participants] | 7 | 7 | 14
Antiarrhythmic [Count of Participants; unit: Participants] | 1 | 1 | 2
Inotropic support prior to enrollment [Count of Participants; unit: Participants] | 2 | 0 | 2
Mechanical Circulatory Support prior to enrollment [Count of Participants; unit: Participants] | 6 | 3 | 9
IABP [Count of Participants; unit: Participants] | 6 | 3 | 9
ACS [Count of Participants; unit: Participants] | 4 | 1 | 5
Acute on Chronic ICM/NICM [Count of Participants; unit: Participants] | 7 | 8 | 15
Mechanical Ventilation [Count of Participants; unit: Participants] | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Episodes of Arrhythmia
Description: requiring intervention (medical therapy or therapy with temporary pacemaker)
Time Frame: up to 96 hours
Measure: Count of Participants; unit: Participants
Groups:
- Control: Patients will receive only standard of care treatment for cardiogenic shock.
Arm/Group | Control | Therapeutic Hypothermia
Number analyzed (Participants) | 10 | 10
Participants | 0 | 1
Statistical Analysis 1: Comparison: Control vs Therapeutic Hypothermia; Test type: Other; p = 1, Fisher Exact

2. Primary Outcome: Number of Participants With Bleeding
Description: requiring transfusions as a direct result of the cooling catheter insertion or secondary to resulting coagulopathy
Time Frame: up to 96 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Therapeutic Hypothermia
Number analyzed (Participants) | 10 | 10
Participants | 0 | 2
Statistical Analysis 1: Comparison: Control Group vs Therapeutic Hypothermia; Test type: Superiority; p = 0.47, Fisher Exact

3. Primary Outcome: Number of Participants With Bloodstream Infection/Suspected Sepsis
Description: confirmed with 2 positive blood cultures or sequential organ failure assessment (SOFA) score >2
Time Frame: up to 96 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Therapeutic Hypothermia
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0
Statistical Analysis 1: Comparison: Control Group vs Therapeutic Hypothermia; Test type: Superiority; p = 1, Fisher Exact

4. Primary Outcome: Number of Participants With Hypokalemia
Description: potassium levels below 3.0mEq/L, not secondary to other identifiable causes
Time Frame: up to 96 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Therapeutic Hypothermia
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0
Statistical Analysis 1: Comparison: Control Group vs Therapeutic Hypothermia; Test type: Superiority; p = 1, Fisher Exact

5. Secondary Outcome: Changes in Cardiac Index
Description: Difference between groups in cardiac index and output
Time Frame: up to 96 hours
Measure: Mean (Inter-Quartile Range); unit: Liter/minute/m^2
Arm/Group | Control Group | Therapeutic Hypothermia
Number analyzed (Participants) | 10 | 10
Liter/minute/m^2 | 2.6 [2.5 to 3.15] | 3.6 [3.1 to 3.9]
Statistical Analysis 1: Comparison: Control Group vs Therapeutic Hypothermia; Test type: Superiority; p = 0.029, Mixed Models Analysis

6. Secondary Outcome: Changes in Systemic Vascular Resistance (SVR)
Description: Mean SVR in population
Time Frame: up to 96 hours
Measure: Mean (Inter-Quartile Range); unit: mm Hg*min/mL
Arm/Group | Control Group | Therapeutic Hypothermia
Number analyzed (Participants) | 10 | 10
mm Hg*min/mL | 965 [891 to 1051] | 702 [667 to 827]
Statistical Analysis 1: Comparison: Control Group vs Therapeutic Hypothermia; Test type: Superiority; p = 0.091, Mixed Models Analysis

7. Secondary Outcome: Cardiac Power Index
Description: Measured 48-96 hours after randomization
Time Frame: up to 96 hours
Measure: Mean (Inter-Quartile Range); unit: W/m^2
Arm/Group | Control Group | Therapeutic Hypothermia
Number analyzed (Participants) | 10 | 10
W/m^2 | 0.61 [0.55 to 0.7] | 0.53 [0.435 to 0.565]
Statistical Analysis 1: Comparison: Control Group vs Therapeutic Hypothermia; Test type: Superiority; p = 0.029, Mixed Models Analysis

8. Secondary Outcome: Cumulative Milrinone Dose
Description: cumulative weight adjusted dosing of milrinone
Time Frame: up to 96 hours
Measure: Mean (Inter-Quartile Range); unit: mg/kg
Arm/Group | Control Group | Therapeutic Hypothermia
Number analyzed (Participants) | 10 | 10
mg/kg | 0.28 [0 to 0.578] | 0.36 [0 to 0.52]
Statistical Analysis 1: Comparison: Control Group vs Therapeutic Hypothermia; Test type: Superiority; p = 0.7, t-test, 2 sided

9. Secondary Outcome: Left Ventricular Ejection Fraction
Description: percent ejection fraction on echocardiogram at 18-24 hours after randomization
Time Frame: up to 18-24 hours
Measure: Mean (Inter-Quartile Range); unit: percent
Arm/Group | Control Group | Therapeutic Hypothermia
Number analyzed (Participants) | 10 | 10
percent | 40.1 [36.2 to 40.8] | 28.1 [22.4 to 62.5]
Statistical Analysis 1: Comparison: Control Group vs Therapeutic Hypothermia; Test type: Superiority; p = 0.516, Fisher Exact

10. Secondary Outcome: All-cause Mortality
Description: All-cause mortality at 90 days was primary outcome/time point of choice.
Time Frame: up to 96 hours, 30 days, and 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Therapeutic Hypothermia
Number analyzed (Participants) | 10 | 10
Participants | 3 | 4
Statistical Analysis 1: Comparison: Control Group vs Therapeutic Hypothermia; Test type: Other; p = 0.75, Kaplan Meier

11. Secondary Outcome: Cumulative Dobutamine Dose
Description: Cumulative dose of weight adjusted dobutamine dobutamine
Time Frame: 96 hours
Population: All trial participants
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Control Group | Therapeutic Hypothermia
Number analyzed (Participants) | 10 | 10
mg/kg | 0 [0 to 1.6] | 0 [0 to 10.75]
Statistical Analysis 1: Comparison: Control Group vs Therapeutic Hypothermia; Test type: Superiority; p = 0.43, t-test, 2 sided

12. Secondary Outcome: Cumulative Dopamine Dose
Description: Cumulative weight adjusted dopamine dose
Time Frame: 96 hours
Population: All patients in study were analyzed
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Control Group | Therapeutic Hypothermia
Number analyzed (Participants) | 10 | 10
mg/kg | 0 [0 to 0.23] | 7.27 [0 to 35.28]
Statistical Analysis 1: Comparison: Control Group vs Therapeutic Hypothermia; Test type: Superiority; p = 0.052, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 90 days
Description: Adverse events were systematically collected and analyzed for these inpatient clinical trial participants. Changes in vitals, clinical condition, need for transfusions, and other events were reported by managing team to trial coordinators. Each relevant event was discussed with the data safety monitoring board.
Arm/Group | Control Group | Therapeutic Hypothermia
All-Cause Mortality (participants affected / at risk) | 3/10 | 4/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 0/10 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=10) | Therapeutic Hypothermia (N=10)
Bradycardic Arrest (General disorders) | 0 (0) | 1 (1) — Patient underwent bradycardia with subsequent PEA arrest during rewarming after cooling. This was classified as a serious adverse event which was deemed to be possibly related to the trial by the Data Safety Monitoring Board (DSMB)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=10) | Therapeutic Hypothermia (N=10)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — 2 patients had mild bleeding with 2-4u transfusion requirements during hospitalization. Both events were deemed as possibly related to trial.
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — Bradycardia during cooling, improved with discontinuation of amiodarone
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1) — Worsening hyperglycemia during cooling in a patient with a history of DM2. Deemed as possibly related to trial.
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) — Patient had hypotension during cooling requiring pressors.
Non-sustained Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — Patient had NSVT after trial enrollment deemed possibly related to the trial
Shivering (General disorders) | 0 (0) | 2 (2) — Shivering related to cooling that was treated with warming blankets and sedation, cessation of cooling was not required
Aspiration Event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient had aspiration during cooling with subsequent concern for sepsis without positive blood cultures. This was classified as a possibly related adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT03141255/Prot_SAP_000.pdf